CLINICAL TRIAL: NCT05437588
Title: Neural-Derived Plasma Exosomal MicroRNAs As Promising Novel Biomarkers for Suicidality and Treatment Outcome in Adolescents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Yogesh Dwivedi, PhD, Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB-300009460; R01MH130539 (NIH)
Record Dates: First submitted 2022-06-23; First posted 2022-06-29 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Major Depressive Disorder; Suicidal Ideas; Suicide, Attempted; MDD; Depression; Depression, Teen; Depression and Suicide; Depression in Adolescence; Suicide
MeSH Terms: conditions — Depressive Disorder, Major; Suicide, Attempted; Depression; Suicide | interventions — Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MDD Participant (Other): Participants with MDD will return at six weeks for a second blood draw and assessments
  Interventions: Genetic: Genetic testing

INTERVENTIONS:
Genetic: Genetic testing — Attempting to identify the genetic biomarker that can identify risk for suicidal ideation and action

SUMMARY:
This study is dedicated to help identify biomarkers for depression and suicide. The purpose of the study is to better understand these links to improve medical and psychiatric care in the future. This research is also to test the effects of standard treatment of depression on improvement in depressive and suicidal behavior and on biomarkers (e.g. miRNA) for these disorders.

ELIGIBILITY:
Inclusion Criteria:

All participants:

1. Physically healthy
2. willing and able to provide informed consent (if under 18 also parent or guardian consent)

MDD participants:

1. A definite diagnosis of DSM-5
2. a Children's Depression Rating Scale-Revised (CDRS-R) score >=30. Suicidal ideation participants: Columbia Suicide Severity Rating Scale (C-SSRS) score >=4 rated over the last two weeks.

Suicide attempt group:

1. Participants will have had an attempt in the previous two weeks that is serious enough to require medical attention and shows evidence of at least a medium level of intent on the Suicide Intent Scale.

Non-psychiatric controls:

1. No history of any major mental illness (excluding specific phobia) or substance use disorder.

Exclusion Criteria:

* Exclusion criteria:

  1. Pregnancy or lactation
  2. post-partum state (being within 2 months of delivery or miscarriage);
  3. homicide risk as determined by clinical interview
  4. any of the following DSM-V diagnoses or categories: a) a lifetime history of psychotic disorder; b) alcohol or drug use disorder (except nicotine/caffeine) within the last month; the use of any hallucinogen (except cannabis), including phencyclidine in the last month; c) bipolar disorder; d) pervasive developmental disorder; e) cognitive disorder; f) DSM-5 paranoid, schizoid, or schizotypal personality disorders (PDs) (participants with other PDs will be allowed as long as MDD criteria are met); g) anorexia nervosa.
  5. recent myocardial infarction or unstable angina, active neoplasm in the past 6 months, immunosuppressive or corticosteroid therapy within the last month, chemotherapy, and head injury or loss of consciousness in the past 6 months
  6. use of hallucinogens (except for cannabis), methamphetamine, or cocaine in the last 2 weeks.

Ages: 10 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2027-06-29 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinical phenotype analysis | 6 Weeks

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UAB Huntsville Regional Medical Campus, Huntsville, Alabama

IPD SHARING:
Plan to Share IPD: Undecided